CLINICAL TRIAL: NCT05174338
Title: Cardiac Amyloidosis Registry Study - A Multi-Center, Longitudinal, Observational Survey of Patients With Cardiac Amyloidosis
Brief Title: Cardiac Amyloidosis Registry Study
Acronym: CARS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Jignesh Patel, MD, PhD, Principal Investigator, Cedars-Sinai Medical Center
Other Study IDs: STUDY00000442
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Amyloidosis, Immunoglobulin Light-chain
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AL and TTR amyloidosis: immunoglobulin light chain amyloidosis (AL) and transthyretin amyloidosis (ATTR)
  Interventions: Other: Registry

INTERVENTIONS:
Other: Registry — Observational, data collection

SUMMARY:
This registry is a observational, multi-center study designed to collect data and analyze it retrospectively on patients with cardiac amyloidosis who have been evaluated and treated at major amyloid centers across the US and internationally between 1997 and 2025.

DETAILED DESCRIPTION:
Amyloidosis is a rare, multisystem disorder in which an insoluble protein is deposited in tissues, leading to organ dysfunction. Several proteins have been identified to potentially lead to amyloid cardiomyopathy (AC). Given the rare nature of these diseases, a large, multi-center effort to describe the characteristics of these patients and their outcomes with novel treatment modalities has not been established. (TBD) academic medical centers from the US and internationally will compile demographic, hemodynamic and organ-involvement data, as well as treatment strategies for AL and TTR amyloidosis.

This registry is an observational, multi-center study designed to collect data and analyze it retrospectively on patients with cardiac amyloidosis who have been evaluated and treated at major amyloid centers across the US and internationally between 1997 and 2025. It is expected that the total patient population will be approximately 5000 patients.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of AL or TTR cardiomyopathy identified or treated within the timeframe
* Specific to CSMC: If the individual provided consent while they were alive, and if sufficient information exists in their chart, their data will be included.
* Information on deceased individuals may be included, but only with the appropriate approval from the external site IRB and/or according to the federal regulations for the protection of human subjects.

Exclusion Criteria:

* At Cedars-Sinai, records that specifically state not to be used in research will not be accessed. Patients who have enacted a No Research Flag or are noted as "Break the Glass" will not be included. For external sites, records that indicate No Research Flag or are noted as "Break the Glass" may be included based on institutional policies and appropriate approvals, as applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Established diagnosis of AL or TTR cardiomyopathy identified or treated
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-01-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Quantify disease severity at diagnosis, progression and survival in patients with cardiac amyloidosis | 1997 - 2025
  Clinical Outcomes: Disease severity at presentation, progression, and survival [time frame 3 years]. Severity and progression determined by change in NYHA Class, NT-ProBNP and troponin.
Quantify incidence of complications from cardiac amyloidosis | 1997 - 2025
  Determine incidence of arrhythmias (atrial fibrillation; ventricular arrhythmias) after diagnosis, renal dysfunction (rise in creatinine and development of end-stage renal disease), stroke, bleeding complications [time frame 3 years]

CONTACTS AND LOCATIONS:
Locations (23):
- United States (22):
  - University of Arizona Sarver Heart Center, Tucson, Arizona
  - UC San Diego Health, Sulpizio Cardiovascular Center, La Jolla, California
  - Scripps Health, La Jolla, California
  - University of California Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - MedStar Health and Vascular Institute/Georgetown University School of Medicine, Washington D.C., District of Columbia
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Weill Cornell Medicine, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - Columbia University Irving Medical Center, Clinical Cardiovascular Research Laboratory for the Elderly (CUMC/CCRLE), New York, New York
  - Duke Health, Durham, North Carolina
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
The study design reflects IPD sharing between researchers based upon agrred set of data elements for study projects in the registry.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available upon entry of IPD into the data base and will remain available for the duration of the study.
Access Criteria: Project participants will have access to IPD only relevant to their approved projects. project approval will be determined collectively by the PIs of all the participating sites.

DOCUMENTS (1):
  • Study Protocol (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT05174338/Prot_002.pdf